CLINICAL TRIAL: NCT00557401
Title: A Multi-Center Randomized, Parallel-Group, Double-Blind, Placebo-Controlled, Study of XP19986 in Subjects With Symptomatic Gastroesophageal Reflux Disease (GERD)
Brief Title: An Efficacy and Safety Study of XP19986 in Subjects With Symptomatic GERD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XP-B-057
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — arbaclofen placarbil; BID protein, human; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- XP19986 SR3, 20 mg QD (Experimental): XP19986, 20 mg QD for approximately 32 days
  Interventions: Drug: XP19986 SR3, 20 mg QD
- XP19986 SR3, 40 mg QD (Experimental): XP19986, 40 mg QD for approximately 32 days
  Interventions: Drug: XP19986 SR3, 40 mg QD
- XP19986 SR3, 60 mg QD (Experimental): XP19986, 60 mg QD for approximately 32 days
  Interventions: Drug: XP19986 SR3, 60 mg QD
- XP19986 SR3, 30 mg BID (Experimental): XP19986, 30 mg BID for approximately 32 days
  Interventions: Drug: XP19986 SR3, 30 mg BID
- Placebo (Placebo Comparator): Placebo for approximately 32 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XP19986 SR3, 20 mg QD — XP19986 Sustained Release (SR) 20 mg tablet taken orally, once daily (QD) for approximately 32 days with titration and taper periods.
  Other Names: arbaclofen placarbil
  Arms: XP19986 SR3, 20 mg QD
Drug: XP19986 SR3, 40 mg QD — XP19986 Sustained Release (SR) 40 mg tablet taken orally, once daily (QD) for approximately 32 days with titration and taper periods.
  Other Names: arbaclofen placarbil
  Arms: XP19986 SR3, 40 mg QD
Drug: XP19986 SR3, 60 mg QD — XP19986 Sustained Release (SR) 60 mg tablet taken orally, once daily (QD) for approximately 32 days with titration and taper periods.
  Other Names: arbaclofen placarbil
  Arms: XP19986 SR3, 60 mg QD
Drug: XP19986 SR3, 30 mg BID — XP19986 Sustained Release (SR) 30 mg tablet taken orally, twice daily (BID) for approximately 32 days with titration and taper periods.
  Other Names: arbaclofen placarbil
  Arms: XP19986 SR3, 30 mg BID
Drug: Placebo — Placebo tablet taken orally for approximately 32 days with titration and taper periods.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
To evaluate efficacy and safety of treatment with XP19986 Sustained Release (SR) Tablet compared to placebo in subjects with symptomatic GERD

ELIGIBILITY:
Inclusion Criteria:

* History and documentation of GERD diagnosed by a gastroenterologist, with symptoms (heartburn and/or regurgitation) on ≥ 3 days during the week prior to screening and prior to randomization

Exclusion Criteria:

* Current or historical endoscopic evidence of erosive esophagitis LA Classification Grade B, C, or D

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Number of heartburn events over the treatment period | 4-weeks

SECONDARY OUTCOMES:
Frequency of regurgitation; severity of heartburn and regurgitation; sleep symptoms | 4-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jay Huff, M.D., Study Director — XenoPort, Inc.
Locations (1):
- MDS Pharma Services, Irvine, California, United States